CLINICAL TRIAL: NCT04937218
Title: Impact Evaluation of GAIN Egg Campaign in Two Nigerian States
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Global Alliance for Improved Nutrition (Other)
Responsible Party: Principal Investigator, Edward Frongillo, Jr., Professor, University of South Carolina
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 101
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Egg Consumption

STUDY DESIGN:
Intervention Model Description: Longitudinal pre- post-evaluation of intervention and comparison group
Who Masked: Outcomes Assessor
Masking Description: Data collectors were masked to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Egg demand creation campaign (Experimental): Egg demand creation campaign using Above-the-line and Below-the-line methods for 14 months. Above-the-line interventions include television, radio, celebrity ambassadors and out-of-home advertising (e.g., billboards). Below-the-line interventions include interpersonal communication activation, trade promotions, point-of-sale materials, food demonstrations and giveaways and door-to-door activation.
  Interventions: Behavioral: Egg demand creation campaign
- Comparison (No Intervention): Comparison arm with no campaign

INTERVENTIONS:
Behavioral: Egg demand creation campaign — Egg demand creation campaign including 14 months of above-the-line and below-the-line messaging.
  Arms: Egg demand creation campaign

SUMMARY:
Improved infant and young child feeding, including dietary quality and diversity, is important for child health and development. In the 2013 Nigeria Demographic and Health Survey, only 18% of children 6-23 months of age received at least 4 food groups in the previous 24 hours. In Kaduna, one of the poorest states, dietary diversity is low and consumption of eggs is infrequent, with households reporting consuming eggs only one day per week. Eggs are a nutrient-dense food, which can contribute enormously to a child's dietary quality. This study evaluates whether a 14-month behavior change intervention about eggs can increase the procurement and consumption of eggs in children 6-59 months of age living in Nigeria. The intervention includes delivery of messages about the health benefits of eggs through Above-the-line methods and Below-the-line methods. The intervention is evaluated using a longitudinal quasi-experimental design in two states in Nigeria with pre- and post-test questionnaires designed to assess changes in acquisition and consumption of eggs.

DETAILED DESCRIPTION:
The Global Alliance for Improved Nutrition (GAIN) seeks to improve dietary quality among children under-five years of age in Kaduna by increasing the demand for eggs through above-the-line and below-the-line behavior change interventions incorporating mass media, social media, and point-of-sale (POS) marketing. Above-the-line (ATL) interventions include television, radio, celebrity ambassadors and out-of-home (OOH) advertising (e.g., billboards). Below-the-line interventions (BTL) include interpersonal communication (IPC) activation, trade promotions, point-of-sale materials, food demonstrations and giveaways and door-to-door activation.

GAIN conducted a quasi-experimental longitudinal study of a demand creation campaign, using ATL and BTL interventions, among families of children 6-59 months of age to determine the impact on egg consumption among children and egg acquisition. Kaduna state was chosen as the intervention arm, and Kano state as the comparison arm. Within Kaduna state, the Kaduna North and Chikun local government areas (LGAs) were selected to receive ATL and BTL demand creation interventions. The comparison state, Kano, received no demand creation campaign.

The principal comparison for measuring the effect of demand creation interventions will be across states, comparing the combined effects of ATL and BTL interventions with the comparison areas which received no intervention.

Investigators also set out to determine the impact of this intervention on mediating outcomes in the hypothesized causal framework. Proximal mediators included caregivers' attitudes and beliefs toward eggs and willingness to pay for eggs.

ELIGIBILITY:
Inclusion Criteria:

* Living in the project areas

Exclusion Criteria:

* Vulnerable families (i.e., families headed by children, homeless families living on the street in the community, families with a severely mentally unstable head of household)

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3453 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Change in the times eggs were consumed by children 6-59 months of age from baseline to endline | From baseline to 14 months
  Change in the average number of times eggs were consumed in the past 7 days from baseline to endline in the two study arms
Change in the consumption of two or more eggs by children 6-59 months of age from baseline to endline | From baseline to 14 months
  Change in the proportion of children consuming at least two eggs in the past 7 days from baseline to endline in the two study arms
Change in the availability of eggs by families of children 6-59 months of age from baseline to endline | From baseline to 14 months
  Change in the proportion of households purchasing eggs and the change in the proportion of households acquiring eggs from baseline to endline in the two study arms

SECONDARY OUTCOMES:
Change in the consumption of any eggs by children 6-59 months from baseline to endline in the two study arms | From baseline to 14 months
  Change in the consumption of one or more eggs by children 6-59 months of age from baseline to endline
Change in caregivers' (of children 6-59 months) attitudes, beliefs, and knowledge of eggs from baseline to endline | From baseline to 14 months
  Change in the mean factor score created from Likert scales of attitudes (attitudes scale, higher score reflects better attitudes towards eggs), perceived benefits (benefits scale, higher score reflects better perceived benefits towards eggs), norms (norms scale, higher score reflects better norms towards eggs), self-efficacy (self-efficacy scale, higher score reflects better self-efficacy), and intention towards eggs (intent to feed eggs to child, higher score reflects more intent to feed eggs) from baseline to endline between the two study arms; change will be examined for a meta factor score combining all scales and each scale separately.
Change in caregivers' willingness to pay for eggs from baseline to endline | From baseline to 14 months
  Change in willingness to pay for eggs, using for example the change in mean maximum price that caregivers would be willing to pay for eggs from baseline to endline between the two study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Frongillo, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of Ibadan, Ibadan, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Reports will be made available. We will provide information on how to make the request to have access to the partial or complete anonymized dataset.
Supporting Information: CSR